CLINICAL TRIAL: NCT05164640
Title: Ischemia in Patients With Non-obstructive Disease (INOCA) in Italy INOCA IT Multicenter Registry"
Acronym: INOCAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Principal Investigator, Chieffo Alaide, Interventional cardiologist, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RF-2019-12369486
Record Dates: First submitted 2021-10-08; First posted 2021-12-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Ischemia
Keywords: non-obstructive coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of coronary physiology (Other): This is a prospective, multicentric, non-randomized , single-arm , open label clinical study.
  Included patients will be studied with invasive functional tests performed during index coronary angiography. These will include FFR, instantaneous Wave-Free Ratio (iFR), Resting Ful-Cycle Ra-tio (RFR), CFR, IMR and provocative Acetylcholine test.
  After the diagnosis of vasospastic angina (VSA) or coronary microvascular dysfunction (CMD) is made, a stratified medical therapy will then be initiated according to the results of physiological assessment according to ESC guidelines and recent EAPCI expert consensus document .
  Interventions: Other: not required

INTERVENTIONS:
Other: not required — This a multicenter, prospective, non-randomized, single-arm, open label clinical study. This design doesn't include control vs intervention arms

SUMMARY:
Prospective, interventional, multicentre, non-randomized, single-arm open-label study that aims to enroll 200 consecutive patients with suspected chronic ischemic heart disease in the absence of obstructive coronary artery disease (INOCA) at clinically indicated coronary angiography in 3 Italian centers.

During coronary angiography, these patients will be simultaneously subjected to a functional and coronary physiology study (according to the methods reported below):

* Functional evaluation with fractional flow reserve (FFR), instantaneous wave-free ratio (iFR), Resting Full-Cycle Ratio (RFR) of angiographic stenosis> 50%;
* In the presence of coronary angiographic stenosis <50% or> 50% but in the presence of a negative functional assessment (FFR> 0.80 and iFR / RFR> 0.90), coronary flow reserve (CFR) and index of microvascular resistance (IMR) will be measured. IMR and CFR will be assessed using intra-coronary guidance;
* In the presence of CFR> 2.0 and IMR <25, tests with acetylcholine will also be performed in order to evaluate the possible presence of epicardial (focal or diffuse) or microvascular spasm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation of chronic ischemic heart disease (IHD), requiring coronary angiography for the diagnosis
* Absence of obstructive CAD at coronary angiography
* Age > 18 years
* Ability to provide a valid informed consent to the study procedure at the time of baseline evaluation

Exclusion Criteria:

* Clinical presentation of acute coronary syndrome (ACS) or cardiogenic shock
* Presence of obstructive CAD with at least 1 significant coronary artery stenosis, defined as diameter stenosis >50% and FFR ≤0.80 (or iFR/RFR ≤0.89)
* Previous coronary artery bypass grafting (CABG)
* Left ventricular systolic dysfunction, defined as ejection fraction (EF) <40%
* Severe valvular heart disease
* Pregnant or breastfeeding women
* Known hypersensitivity or contraindication to any of the drugs used for coronary physiology testing (adenosine, nitrates, acetylcholine)
* Inability or unwillingness to provide a valid informed consent to the study procedure at the time of baseline evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
investigate the prevalence of INOCA in women vs. men | 3 year
  1. To investigate the prevalence of INOCA in women vs. men who are referred for a clinically indicated coronary angiography in three Centers in North-ern, Central and Southern Italy;
stratify in INOCA endotypes patients | 1 day (during physiology tests)
  2. to stratify in INOCA endotypes patients according to the presence or absence of alternative (i.e. non obstructive CAD) causes of myocardial ischemia detected during CA clinically indicated through physiology tests
implement a stratified therapy | 1 year
  3. to implement a stratified therapy in these patients considering the different INOCA endotypes and evaluate the impact on angina class and quality of life as well as cardiac hospitalization and coronary revascularization during 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alaide Chieffo, MD, Principal Investigator — IRCCS San Raffaele
Locations (3):
- Italy (3):
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliera Universitaria Federico II,, Napoli
  - Fondazione Policlinico Universitario A. Gemelli IRCCS,, Roma

IPD SHARING:
Plan to Share IPD: No